CLINICAL TRIAL: NCT05753215
Title: Omadacycline Versus Standard-of-Care Oral Antibiotic Treatment for Bone and Joint Infections: An Open-Label, Non- Inferiority, Randomized, Controlled Trial
Brief Title: Controlled Trial of Omadacycline Randomized Treatment Given for Bone and Joint Infection
Acronym: CORGI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Chapman University (Other); Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Principal Investigator, loren g miller, Chief, Division of Infectious Diseases, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22885-01
Record Dates: First submitted 2023-02-03; First posted 2023-03-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bone Infection; Joint Infection; Bone and Joint Infection
MeSH Terms: interventions — omadacycline; Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects will receive an omadacycline-containing regimen versus SOC. Prior to randomization, SOC antibacterial therapy will be selected by the subject's treating physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- omadacycline (Experimental): Omadacycline will be administered 300 mg orally daily without the loading dose. We chose to omit the loading dose given that many of the enrolled subjects would have received an IV therapy prior to omadacycline initiation and notable gastrointestinal intolerabilities (nausea/vomiting) based on Phase-3 trial data. Subjects receiving omadacycline will be counseled on appropriate timing of administration (fast for 4 hours before dosing and no food for 2 hours after dosing) in light of the known food effects on drug absorption. They will be instructed to avoid use of products containing aluminum, calcium, or magnesium, bismuth subsalicylate, and iron containing preparations such as dairy, antacids, and multivitamins for 4 hours post-dosing.
  Interventions: Drug: Omadacycline Pill
- standard of care antibiotic (Other): Standard of care as determined by primary care team
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Omadacycline Pill — Omadacycline will be administered 300 mg orally daily without the loading dose.
  Other Names: nuzyra
  Arms: omadacycline
Drug: Standard of Care — Prior to randomization, SOC antibacterial therapy will be selected by the subject's treating physician.
  Arms: standard of care antibiotic

SUMMARY:
The study design is a randomized, open-label, clinical trial of omadacycline vs Standard of Care (SOC) antibiotics for bone and join infection (BJI) treatment. Study participants will have their BJI regimen chosen by their treating physicians, (typically Infectious Diseases for hardware and prosthetic joint infections, or multidisciplinary Limb Salvage team for diabetic foot infections) prior to enrollment. Then participants will be randomized to an omadacycline-containing regimen versus the a priori chosen SOC regimen. Participants must require between 4 and 12 weeks of therapy for their BJI. The exact duration of therapy will be decided by the participants' treating physician. At 12 weeks, if the treating physician wishes to extend therapy, participants receiving omadacycline will be transitioned to other SOC antibiotics.

Once enrolled, participants will be followed via in-person clinic visits at the following intervals: weeks 0, 2, 4, 8, and 12. A final in-person visit will occur 2 weeks post-treatment completion. A phone survey will occur 3 months post-treatment completion. Participants in the SOC group will follow the same schedule.

Oral once-daily dosing options for S. aureus and Coagulase negative Staphylococcus are essentially non-existent. Thus, omadacycline possesses a novel and advantageous option for BJI treatment. Its convenient dosing regimen will almost certainly be associated with improved adherence, and higher adherence may, in turn, improve clinical outcome. Investigators hypothesize that omadacycline will be a well-tolerated and efficacious oral antibiotic for BJIs and will be associated with improved adherence compared with standard of care oral antibiotics. Investigators believe omadacycline addresses the unmet need for an oral antibiotic that is well-tolerated and efficacious for use as a prolonged therapy for BJIs. To this aim, investigators will perform a randomized, open-label clinical trial of omadacycline to SOC antibiotics for BJIs.

DETAILED DESCRIPTION:
The design of this study is a prospective, open-label, randomized clinical trial of omadacycline vs SOC antibiotics for the treatment of BJIs. We will follow subjects for between 16 and 24 weeks, depending on the length of their antibiotic treatment, for the purpose of determining tolerability, safety, and treatment success of prolonged use (> 4 weeks) of omadacycline in the treatment of BJIs. Subjects will be enrolled regardless of race, ethnicity, or gender (as long as they are within 18 - 85 years of age).

Subjects will be given omadacycline-containing regimen versus SOC. Omadacycline will be administered 300 mg orally daily without loading dose duration of therapy of between 4 and 12 weeks. The exact duration of therapy will be decided by the subject's treating physician. In other words, the primary/consulting physician who is managing the treatment of the subject's bone and joint infection will be the one who decides the length of the antibiotic treatment.

Safety and tolerability of omadacycline through this study will be guaranteed for 12 weeks. At 12 weeks, if the treating physician wishes to extend therapy, subjects receiving omadacycline will be transitioned to other SOC antibiotics. Medications will be provided by the Investigational Drug Service (IDS) on The Lundquist Institute/Harbor-UCLA campus, which supplies all research related medications to study subjects at our center.

Subjects will be enrolled as outpatients or as inpatients when discharge is expected in the near future (< 1 week). Drs. Loren Miller and/or Amy Kang, the Co-Principal Investigators, will advise the hospital staff of the study and seek their assistance in identifying and notifying the study staff of possible subjects who have presented to the Emergency Department, inpatient units, or outpatient clinic with BJI.

Our primary endpoint is treatment success 2-weeks after therapy completion. We hypothesize that omadacycline will be non-inferior to SOC antibiotics for BJI treatment. For descriptive purposes, treatment outcome will be further sub-categorized as one of the following outcomes: treatment success, failure due (or probably due) to medication, and failure not due (or unlikely due) to medication (e.g., surgical issues such as inadequate source control). For our primary analysis, we will dichotomize outcomes to treatment success and treatment failure. Treatment success will be defined as the lack of definite treatment failure. Treatment failure will be defined using the definition utilized in the OVIVA trial. Specifically, definite failure will be defined as the presence of at least one clinical criterion (draining sinus tract arising from bone or prosthesis or the presence of frank pus adjacent to bone or prosthesis), microbiologic criterion (phenotypically indistinguishable bacteria isolated from two or more deep-tissue samples or a pathogenic organism from a single closed aspirate or biopsy), or histologic criterion (presence of characteristic inflammatory infiltrate or microorganisms).

For descriptive purposes, treatment failure will be subdivided into definite, probable, and possible failure. Using definitions from the OVIVA trial, definite treatment failure will be defined by one or more of the following: a) isolating bacteria from 2 or more samples of bone/peri-prosthetic tissue, where the bacteria isolated from these samples were indistinguishable according to routine laboratory tests, including the antibiogram; b) a pathogenic organism (e.g. Staphylococcus aureus but not Staphylococcus epidermidis) on a single, closed, biopsy of native bone or periprosthetic tissue; c) diagnostic histology on bone/peri-prosthetic tissue; d) a draining sinus tract arising from bone/prosthesis; or e) frank pus adjacent to bone/ prosthesis. If any of these criteria are met, then the category "definitive" infection will be applied. Where these criteria are not met, the following criteria will be used to determine "probable" or "possible" infection: Infection will be categorized as "probable" where microbiological sampling had not been undertaken, AND none of the other criteria for definite infection had been fulfilled AND any one of the following are met: a) Radiological or operative findings of periosteal changes suggesting chronic osteomyelitis OR b) Radiological findings suggesting vertebral infection OR c) The development of a discharging wound after an orthopedic procedure where prosthetic material had been implanted OR d) The presence of deep pus close to but not adjacent to bone/prosthetic joint/orthopedic device OR e) The presence of peri-prosthetic necrotic bone OR f) Rapid loosening of a joint prosthesis/orthopedic device (i.e. leading to localized pain in less than 3 months since implantation) in the absence of a mechanical explanation for rapid loosening. Infection will be categorized as "possible" where microbiological sampling had been undertaken with negative results (according to criteria described above for "definite" infection) AND other criteria for definite infection were not fulfilled AND in addition one or more of the criteria listed a) to f) above is met.

Secondary endpoints include treatment success, defined as lack of any category of treatment failures (definite, probable, and possible) two weeks after therapy completion, long-term treatment success, defined as lack of definite treatment failures 3 months after treatment completion, long-term safety and tolerability, and medication adherence. We will measure long-term treatment success by performing a phone survey 3 months after antibiotic completion. Medication adherence will be measured by self-report. Unplanned surgical procedures prompted by inadequate infection control will be categorized as treatment failure. Recurrence of signs or symptoms of BJIs after resolution will be considered a long-term treatment failure.

Subjects will receive an omadacycline-containing regimen versus SOC. Prior to randomization, SOC antibacterial therapy will be selected by the subject's treating physician. Omadacycline will be administered 300 mg orally daily without the loading dose. We chose to omit the loading dose given that many of the enrolled subjects would have received an IV therapy prior to omadacycline initiation and notable gastrointestinal intolerabilities (nausea/vomiting) based on Phase-3 trial data. Subjects receiving omadacycline will be counseled on appropriate timing of administration (fast for 4 hours before dosing and no food for 2 hours after dosing) in light of the known food effects on drug absorption. They will be instructed to avoid use of products containing aluminum, calcium, or magnesium, bismuth subsalicylate, and iron containing preparations such as dairy, antacids, and multivitamins for 4 hours post-dosing. Of note, omadacycline is intrinsically resistant to Pseudomonas, Proteus, Providencia, and Morganella. If any of these organisms are isolated and considered to be clinically relevant at the treating physician's discretion, subject will receive concomitant oral or IV antibiotics in addition to omadacycline. In the SOC group, oral therapy is required for S. aureus treatment; adjunctive IV antibiotics will be permitted, similar to the omadacycline arm.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of BJI or probable BJI as defined clinically using radiologic (e.g., MRI), surgical (e.g., intra-operative findings), and/or clinical (e.g., probe to bone) definitions
2. BJI caused by or suspected to be caused by organisms that omadacycline is expected to be active against
3. Planned treatment duration of 4-12 weeks
4. Plans to continue or initiate treatment in outpatient setting
5. Age 18-85
6. Limited planned course of antibiotics (i.e., no indefinite treatment plans for chronic suppression)
7. Able to take oral medications
8. Able to come to the research clinic for study follow-up visits for the study period
9. If a woman is of childbearing potential, she must consistently use two acceptable methods of contraception (IUD, injectable contraceptive, birth control patch, OCP, barrier method, abstinence) from baseline through the course of antibiotics (4-12 weeks). If a male patient's sexual partner is of childbearing potential, the male patient must acknowledge that they will consistently use an acceptable method of contraception as defined above from baseline through the course of antibiotics (4-12 weeks)

Exclusion Criteria:

1. Pregnancy or breast feeding. Women of childbearing potential must have a negative urine or serum pregnancy test result within 1 day prior to initiation of study drug
2. Hypersensitivity to tetracycline-class antibiotics
3. BJI caused by fungi or mycobacteria
4. BJI complicated by endocarditis, central nervous system involvement such as subdural abscess, or any foci of metastatic infection, such as renal or splenic abscesses
5. Prosthetic joint infections that have not undergone both stages of two stages of surgical treatments (i.e., subjects are only eligible after the 2nd stage surgery has been completed and typically 6 weeks of IV therapy has been completed)
6. Hematogenous BJI prior to adequate treatment for bacteremia (i.e., subjects are only eligible after adequate IV course of bacteremia is completed and additional oral therapy is still required for infection "mop up")
7. Any medical, psychological, or social condition that, in the opinion of the Investigator, would prevent the patient from fully participating in the study or would represent a concern for study compliance or constitute a safety concern to the patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To compare the treatment success, as defined by lack of definite treatment failure, of omadacycline versus standard of care (SOC) antibiotics for bone and joint infections (BJIs) two weeks after therapy completion. | 2 weeks post-therapy
  We will dichotomize outcomes to treatment success and treatment failure. Treatment success will be defined as the lack of definite treatment failure. Treatment failure will be defined using the definition utilized in the OVIVA trial. Specifically, failure will be defined as the presence of at least one clinical criterion (draining sinus tract arising from bone or prosthesis or the presence of frank pus adjacent to bone or prosthesis), microbiologic criterion (phenotypically indistinguishable bacteria isolated from two or more deep-tissue samples or a pathogenic organism from a single closed aspirate or biopsy), or histologic criterion (presence of characteristic inflammatory infiltrate or microorganisms).

SECONDARY OUTCOMES:
Quantify the long term efficacy of omadacycline for BJIs, both non-hardware and hardware associated after therapy completion. | 3 months post-therapy
  We will measure long-term efficacy by performing a phone survey 3 months after antibiotic completion. Definition of treatment efficacy will be same as primary endpoint. Unplanned surgical procedures prompted by inadequate infection control will be categorized as treatment failure. Recurrence of signs or symptoms of BJIs after resolution will be considered a long-term treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Loren G. Miller, MD, MPH, Principal Investigator — The Lundquist Institute For Biomedical Innovation at Harbor-UCLA Medical Center; Amy Y. Kang, PharmD, BCIDP, Principal Investigator — Chapman Univeristy
Locations (1):
- The Lundquist Institute For Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No